CLINICAL TRIAL: NCT04068467
Title: Evaluation of mHealth for Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Dror Ben-Zeev, Professor, School of Medicine: Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00006898
Record Dates: First submitted 2019-08-07; First posted 2019-08-28 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Major Depressive Disorder; Bipolar Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Mobile Application; SMI; EHealth; E-Health; Health Technology; mHealth; m-Health; Mobile Health; Serious Mental Illness; Electronic Health
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Instructed to download the app and use the app daily for 30 days.
  Interventions: Other: Smartphone App
- Waitlist Control (Active Comparator): Waitlist control.
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Other: Smartphone App — The application consists of content areas focused on mental health.
  Arms: Active
Other: Waitlist Control — Waitlist control
  Arms: Waitlist Control

SUMMARY:
This study is a waitlist control trial evaluating the acceptability and preliminary efficacy of a smartphone application with people with mental illness.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Owns an Android or iPhone smartphone with WiFi or 3G/4G capabilities (required for data transmission)
* Has diagnosis of Schizophrenia, Schizoaffective Disorder, Bipolar Disorder or Major Depression
* English speaker

Exclusion Criteria:

* Does not live in the U.S.
* Has already participated in the study
* Unavailable for 60 days
* Currently incarcerated or hospitalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Depressive Symptoms | Baseline, 30 days, 60 days
  The Beck Depression Inventory is a self-reported 21-item inventory, scores range from 0-63 and items are summed to compute the total score. A higher score represents more depressive symptoms.
Change in Paranoid Thinking | Baseline, 30 days, 60 days
  The Green Paranoid Thoughts Scale Parts A & B is a 32-item scale, the total score is summed with a range of 16-80. A higher score represents more symptoms of paranoid thinking.
Change in Anxiety Symptoms | Baseline, 30 days, 60 days
  The Generalized Anxiety Disorder 7-item Scale is summed with a total score range of 0-21. Higher scores represent more symptoms of anxiety.
Change in Psychotic Symptoms | Baseline, 30 days, 60 days
  The Hamilton Program for Schizophrenia Voices Questionnaire is a 13-item questionnaire, 9 of the items are scored 0 (least severe or impairing) to 4 (most severe). The total score is intended to indicate the overall severity of psychotic symptoms. Total score range is 0-36. The remaining 4 items are intended to assess qualitative aspects.
Participant Acceptability | 30 days
  Participant Acceptability/Usability Ratings Scale is a 26-item scale measuring participant-rated acceptability of the intervention. Participants rate statements on a scale of Disagree (0), Neutral (1), or Agree (2). Items are summed to create a total score and a higher total score indicates greater acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Dror Ben-Zeev, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Ben-Zeev D, Chander A, Tauscher J, Buck B, Nepal S, Campbell A, Doron G. A Smartphone Intervention for People With Serious Mental Illness: Fully Remote Randomized Controlled Trial of CORE. J Med Internet Res. 2021 Nov 12;23(11):e29201. doi: 10.2196/29201. PMID 34766913